CLINICAL TRIAL: NCT02633852
Title: A 12-month, Multicenter Study to Evaluate the Efficacy of Treat and Extend Regimen (TER) of Aflibercept (EYLEA) 2mg /0.05 ml as a Second Line Treatment for Diabetic Macular Edema
Brief Title: Multicenter Study to Evaluate the Efficacy of Treat and Extend Regimen of Aflibercept (EYLEA) as a Second Line Treatment for Diabetic Macular Edema
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHOTADI- HMO-CTIL
Record Dates: First submitted 2015-11-25; First posted 2015-12-17 (Estimated); Last update posted 2018-09-14 (Actual); Status verified 2017-09

CONDITIONS: Diabetic Macular Edema (DME)
Keywords: Diabetic Macular Edema (DME); Aflibercept (EYLEA)
MeSH Terms: interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Aflibercept (EYLEA) 2mg /0.05 ml (Experimental): Aflibercept (EYLEA) 2mg /0.05 ml
  Interventions: Drug: Aflibercept

INTERVENTIONS:
Drug: Aflibercept
  Other Names: EYLEA

SUMMARY:
A 12-month, Multicenter Study to Evaluate the Efficacy of Treat and Extend Regimen (TER) of Aflibercept (EYLEA) 2mg /0.05 ml as a Second Line Treatment for Diabetic Macular Edema - TADI Study

DETAILED DESCRIPTION:
A prospective, multicenter, single arm study. The study group will be composed of both type 1 or 2 diabetes mellitus patients with center involving DME. Patients with partial or incomplete response to first-line Bevacizumab (Avastin) treatment of at least 4 monthly intravitreal injections and no longer than 12 months of treatment (maximum 12 injections ) the last 3 injections must be up to 4-6 weeks . Only one eye of each patients can be recruited to the study (fellow eye will receive standard of care treatment).

The study eye will receive intravitreal injection of aflibercept 2mg/0.05ml at enrolment (day 0). The next follow up visit will be 4 weeks later. At any visit, if sub- or intra-retinal (or both) fluid is present or if central macular sub-field thickness according to SD-OCT of larger than 300 micron (Heidelberg Spectralis OCT or equivalent), the patient will receive intravitreal injection of aflibercept 2mg/0.05ml and treatment interval will remain 4 weeks. In case that there will not be resolution or improvement (define as decrease in central macular sub-field thickness of 10% or more from the previous visit or gain of one ETDRS line or more), the intravitreal injection of aflibercept will be discontinued after 6 monthly injections and the patient will be followed every 4 weeks. If there will be worsening of 10% or more in macular thickness and/or loss of one EDTRS line or more of acuity following treatment discontinuation then injections will be resumed. In cases when there will be no sub- or intra-retinal fluid on OCT 4 weeks after an injections, a treat and extend regimen (TER) will be applied.

At any time point there is an option for rescue treatment if there will be worsening of more than 10% or increase of 50 micron in macular thickness and loss of one EDTRS line (5 letters) or more of acuity, or per the decision of the investigator.

Patients will receive injection of aflibercept 2mg/0.05ml, and the follow up interval will be extended by2 weeks. Maximal treatment interval will be 12 weeks . At any point where sub- or intra-retinal (or both) fluid will appear after the TER regimen was initiated, the interval between visits and treatments will be reduced back to previous interval which obtained a fluid free macula. The follow up period will be 52 weeks.

After 6 months, focal laser phothocoagulation can be added if needed.

ELIGIBILITY:
Inclusion Criteria:

Ophthalmic Inclusion Criteria

1. Incomplete response to previous intravitreal treatment, defined as remaining of sub or intraretinal (or both) fluid involving the fovea per OCT after at least 6 monthly intravitreal injections and no more than 18 months of treatment (maximum 18 intravitreal injections). The last 3 injections must be up to 4-6 weeks apart. The interval from last treatment to day 0 treatment of the study should be up to 6 months. If there will be 10% or more of improvement in central macular sub-field thickness according to SD-OCT, in screening compared with examination 4-6 weeks following last bevacizumab injection patient cannot be recruited to the study. Patients that will have an increase in central thickness of more than 50 microns following 3 intravitreal injections will be allowed to participate in the study without the required need of 6 intravitreal injections.
2. Central macular sub-field thickness according to SD-OCT of at least 300 micron (Heidelberg Spectralis OCT or equivalent).
3. Best corrected visual acuity in the study eye 20/200 and better, .
4. Clear ocular media and adequate pupillary dilatation to allow fundus imaging.
5. Intraocular pressure (IOP) of 21 mmHg or less.

Exclusion Criteria:

Ophthalmic Exclusion Criteria

1. An ocular condition is present such that, in the opinion of the investigator, visual acuity loss would not improve from resolution of macular edema (e.g., foveal atrophy, pigmentabnormalities, dense sub-foveal hard exudates).
2. An ocular condition is present (other than diabetes) that, in the opinion of the investigator, might affect macular edema or alter visual acuity during the course of the study (e.g., vein occlusion, uveitis or other ocular inflammatory disease, neovascular glaucoma, etc.).
3. History of pan-retinal photocoagulation or focal laser treatment within three months prior to enrollment or anticipated need for pan-retinal photocoagulation in the six months following enrollment.
4. History of intraocular surgery (including vitrectomy, cataract extraction, scleral buckle, any intraocular surgery, etc.) within prior three months or anticipated within the next six months following enrollment.

General Exclusion Criteria

1. Significant renal disease, defined as a history of chronic renal failure requiring dialysis or kidney transplant.
2. A condition that, in the opinion of the investigator, would preclude participation in the study (e.g., unstable medical status including blood pressure, cardiovascular disease, and glycemic control).
3. Any treatment with an investigational agent in the 60 days prior to trial entry for any condition.
4. Known serious allergies to the fluorescein dye used in angiography (mild allergy amenable to treatment is allowable), or to the components of the aflibercept formulation.
5. For women of child-bearing potential: pregnant or lactating or intending to become pregnant within the next 24 months.Women who are potential study participants should be questioned about the potential for pregnancy. Investigator judgment is used to determine when a pregnancy test is needed.
6. Stroke or Myocardial infraction within 6 months of trial entry. -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2016-05-24 (Actual); Primary Completion 2018-08-28 (Actual); Study Completion 2018-09-06 (Actual)

PRIMARY OUTCOMES:
macular thickness changes | At week 52
  Assess macular thickness changes following second line therapy with aflibercept using treat-and-extend algorithm

SECONDARY OUTCOMES:
visual acuity | At week 52
  Evaluate the change in visual acuity
treatment/injection number required | At week 52
  Assess treatment/injection number required
progression of diabetic retinopathy | At week 52
  Assess progression of diabetic retinopathy